CLINICAL TRIAL: NCT01333059
Title: A Randomized, Double-blind, Controlled Trial of Cycling Continuous Sedative Infusions in Critically Ill Pediatric Patients Requiring Mechanical Ventilation
Brief Title: Cycling of Sedative Infusions in Critically Ill Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to adequately enroll over a reasonable enrollment period.
Sponsor: Javier Gelvez, MD (Other)
Responsible Party: Sponsor-Investigator, Javier Gelvez, MD, M.D., Cook Children's Health Care System
Organization: Cook Children's Health Care System (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sedation Cycling
Record Dates: First submitted 2011-04-06; First posted 2011-04-11 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Failure
Keywords: Sedation; Cycling; Pediatric
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Midazolam; Saline Solution; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): In this arm Fentanyl and Midazolam was replaced with placebo (normal saline) during cycling.
  At cycling time for midazolam, the continuous infusion of midazolam was stopped by the bedside nurse. The nurse started a pump containing a syringe labeled "Study Drug M" which contained the placebo drug (normal saline). The switch to Study Drug M occurred twice daily at 0800 and 2000 for a period of 3 hours each. At cycling time for fentanyl, the continuous infusion of fentanyl was stopped by the bedside nurse. The pump containing a syringe labeled "Study Drug F," which contained the placebo drug (normal saline), was started. The switch Study Drug F occurred twice daily at 1400 and 0200 for a period of 3 hours each.
  Dosing was done per standard of care and not prescribed per protocol
  Interventions: Drug: Midazolam; Drug: Normal saline; Drug: Fentanyl
- Control Group (Active Comparator): In this arm, midazolam and fentanyl were administered during cycling.
  At cycling time for midazolam, the continuous infusion of midazolam was stopped by the bedside nurse. The nurse started a pump containing a syringe labeled "Study Drug M" which contained the control drug (midazolam). The switch to Study Drug M occurred twice daily at 0800 and 2000 for a period of 3 hours each. At cycling time for fentanyl, the continuous infusion of fentanyl was stopped by the bedside nurse. The pump containing a syringe labeled "Study Drug F," which contained the control drug (fentanyl), was started. The switch to Study Drug F occurred twice daily at 1400 and 0200 for a period of 3 hours each.
  Dosing was done per standard of care and not prescribed per protocol.
  Interventions: Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Midazolam
  Other Names: Versed, Study Drug M
Drug: Normal saline
  Other Names: Placebo
  Arms: Experimental Group
Drug: Fentanyl
  Other Names: Subsys, Duragesic, Abstral, Lazanda, IONSYS, Study Drug F

SUMMARY:
The purpose of this study is to determine if the reduction of the total amount of sedative critically pediatric ill patients receive in the PICU will achieve a significant decrease in mechanical ventilation days and a decrease in the overall length of stay in the PICU and hospital.

DETAILED DESCRIPTION:
Continuous sedative infusions have been associated with longer duration of mechanical ventilation, longer stay in the intensive care unit (PICU) and total hospital stay. Also, extended duration of continuous sedative infusions limits the ability to assess for adequate neurologic function.

There is, however, no published data on the use of daily interruption of continuous sedative infusions in pediatric patients, nor are there any recommendations from the leading pediatric critical care groups regarding this issue. Infants and children exposed to noxious stimuli (endotracheal tube, endotracheal suctioning, mechanical ventilation, indwelling catheters) in addition to an unknown environment are less likely to cooperate during normal daily interventions in the PICU. Continuous infusions of benzodiazepines and opioids in addition to as needed (PRN) bolus doses have been the standard of care in our institution for mechanically ventilated patients.

The study seeks to determine if reducing the total dose of sedatives, by holding them in a cyclical manner, will be a safe and effective intervention that will not increase adverse patient outcomes. This will be achieved by limiting the patient tolerance to the sedatives, decreasing the body total deposit of sedatives and subsequently decreases awakening time when patient is ready for extubation.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 18 years of age
* Intubated and mechanically ventilated
* Expected to require continuous infusions of sedatives for at least 48 hours
* Parent or legal guardian available for informed consent
* Males and females of any race are eligible

Exclusion Criteria:

* Less than 72 hours after surgery
* Cyanotic heart disease with unrepaired or palliated right to left intracardiac shunt
* Critical airway (according to PICU Attending)
* Ventilator dependent (including noninvasive) on PICU admission
* Greater than 48 hours of continuous sedation infusion(s)
* Neuromuscular respiratory failure
* Managed by patient controlled analgesia (PCA) or epidural catheter
* Known allergy to any of the study medications (fentanyl or midazolam)
* Family/Medical team have decided not to provide full support (patient treatment considered futile)
* Patient requires ECMO
* Head trauma requiring intracranial pressure monitoring
* Pregnancy
* Following resuscitation from cardiorespiratory arrest whose initial pH is < 6.9
* ICU Attending judgment that patient should be excluded for safety reasons

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gelvez, MD, Principal Investigator — Cook Children's Physician Network; Linda L Thompson, MD, Principal Investigator — Cook Children's Physician Network
Locations (1):
- Cook Children's Medical Center, Fort Worth, Texas, United States

REFERENCES:
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Ista E, van Dijk M, Tibboel D, de Hoog M. Assessment of sedation levels in pediatric intensive care patients can be improved by using the COMFORT "behavior" scale. Pediatr Crit Care Med. 2005 Jan;6(1):58-63. doi: 10.1097/01.PCC.0000149318.40279.1A. PMID 15636661
- [Background] van Dijk M, Peters JW, van Deventer P, Tibboel D. The COMFORT Behavior Scale: a tool for assessing pain and sedation in infants. Am J Nurs. 2005 Jan;105(1):33-6. doi: 10.1097/00000446-200501000-00019. No abstract available. PMID 15659992
- [Background] Kress JP, Gehlbach B, Lacy M, Pliskin N, Pohlman AS, Hall JB. The long-term psychological effects of daily sedative interruption on critically ill patients. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1457-61. doi: 10.1164/rccm.200303-455OC. Epub 2003 Oct 2. PMID 14525802
- [Background] Kress JP, Vinayak AG, Levitt J, Schweickert WD, Gehlbach BK, Zimmerman F, Pohlman AS, Hall JB. Daily sedative interruption in mechanically ventilated patients at risk for coronary artery disease. Crit Care Med. 2007 Feb;35(2):365-71. doi: 10.1097/01.CCM.0000254334.46406.B3. PMID 17205005
- [Background] Colville G, Kerry S, Pierce C. Children's factual and delusional memories of intensive care. Am J Respir Crit Care Med. 2008 May 1;177(9):976-82. doi: 10.1164/rccm.200706-857OC. Epub 2008 Jan 31. PMID 18244955
- [Background] Connolly D, McClowry S, Hayman L, Mahony L, Artman M. Posttraumatic stress disorder in children after cardiac surgery. J Pediatr. 2004 Apr;144(4):480-4. doi: 10.1016/j.jpeds.2003.12.048. PMID 15069396
- See also: Click here for more information about this study: A randomized, double-blind, controlled trial of cycling continuous sedative infusions in critically ill pediatric patients requiring mechanical ventilation — http://www.cookchildrens.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 14 | 11
Completed | 8 | 8
Not Completed | 6 | 3
Not completed — Physician Decision | 3 | 3
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 11 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 0.24 [0.05 to 3.03] | .20 [0.04 to 17.31] | 0.22 [0.04 to 17.31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 6 | 5 | 11
  Race/Ethnicity: Hispanic or Latino | 6 | 6 | 12
  Race/Ethnicity: African American | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Duration of Mechanical Ventilation Days
Description: Participants will be followed for an expected average of 4 days. The Data Safety Monitoring Group will review the data every 6 months.
Time Frame: From date of randomization until the date of discharge from PICU, assessed up to 1 month
Population: In October of 2012, the DSMB unanimously voted to close this study due to safety concerns and inactivity. The Board noted that recruitment goals had not been met and statistical analysis could not be made with current data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 14 | 11
days | 10.14 (5.55) | 5.82 (1.85)

2. Secondary Outcome: PICU Length of Stay
Description: Participants will be followed for an expected average of 7 days. This secondary endpoint is to be evaluated every six months.
Time Frame: From date of randomization until the date of discharge from PICU, assessed up to 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 14 | 11
days | 13.93 (7.49) | 9.82 (6.75)

3. Secondary Outcome: Hospital Length of Stay
Description: Participants will be followed for an expected average of 7 days in PICU and 10 days of hospitalization. This secondary endpoint is to be evaluated every six months.
Time Frame: From date of hospital admission to date of hospital discharge, assessed up to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 14 | 11
days | 25.21 (16.69) | 20.82 (17.80)

ADVERSE EVENTS:
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/11
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/11
Other Adverse Events (participants affected / at risk) | 7/14 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=14) | Control Group (N=11)
Graft vs Host Disease (Immune system disorders) | 0 (0) | 1 (1) — Unrelated
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0) — Unrelated: required ECMO intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=14) | Control Group (N=11)
FiO2 increased (Surgical and medical procedures) | 7 (8) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes